CLINICAL TRIAL: NCT06815913
Title: To Develop and Introduce Into Polyclinic Practice a Register of Patients with Experience of Myocardial Infarction and Acute Cerebrovascular Disease
Status: Active, not recruiting | Type: Observational
Sponsor: State Institution "Republican Scientific and Practical Center" Cardiology, Belarus (Other)
Responsible Party: Principal Investigator, Pabivantsava Natallia, Head of the Laboratories of Comorbid Cardiology, RSPC Cardiology, Ph.D (Medicine), State Institution "Republican Scientific and Practical Center" Cardiology, Belarus
Other Study IDs: 2161/29590637
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction (MI); Acute Cardiovascular Disease
Keywords: registry; multimorbidity; chronic non-communicable diseases; cardiovascular diseases; myocardial infarction; acute cerebrovascular disease
MeSH Terms: conditions — Myocardial Infarction; Noncommunicable Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- myocardial infarction: Some patients with non-fatal myocardial infarction
- acute cerebrovascular disease: Hospitalization due to cardiovascular diseases, some patients with hospitalization due to cardiovascular diseases

SUMMARY:
This is a retrospective observational study using the methodology of creating medical registries. The expected number of patients included in the registry is about 2000 patients with myocardial infarction and/or ACVD of any duration and concomitant non-cardiac diseases of therapeutic profile in pilot healthcare organizations for any reason during 2019-2022 based on the source medical records data.

DETAILED DESCRIPTION:
The implementation of the task results will improve the efficiency of secondary and tertiary prevention of diseases of the circulatory system - pathology that makes the greatest contribution to the main medical-demographic and socio-economic losses of the state by determining the number of groups with the highest risk of death in outpatient and polyclinic institutions among patients after myocardial infarction, ACVD, living in the Republic of Belarus, to create programs of additional measures to reduce morbidity and mortality of the population based on a comparison of register data and official statistical forms, which will ultimately affect the reduction in the incidence of non-fatal recurrent cardiovascular events in individuals after AMI, ACVD and / or their combination of any duration in the range of 0.2-1% of the indicators determined during the study.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who applied to the pilot ambulatory health care organizations between 2019-2022 in order to identify and "look for" patients after acute cardiovascular event, but who were not monitored for that event for various reasons (statute of limitations, refusal, relocation, etc.);
2. All patients discharged from hospitals with a final diagnosis of AMI/ACVD, assigned territorially to the pilot polyclinics in the period 2019-2022.
3. Presence of a history of AMI and/or ACVD;
4. Age 18 years and older.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who applied to the pilot ambulatory health care organizations between 2019-2022 in order to identify and "look for" patients after acute cardiovascular event, but who were not monitored for that event for various reasons (statute of limitations, refusal, relocation, etc.); meeting the inclusion criteria and not meeting the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality from other causes | 3 years
  number of deaths from other diseases

OTHER OUTCOMES:
Time to combined end point | 3 years
  non-fatal myocardial infarction or non-fatal cerebral stroke or coronary/carotid revascularization
Proportion of patients with non-fatal myocardial infarction | 3 years
  non-fatal myocardial infarction
Proportion of patients with non-fatal cerebral stroke | 3 years
  non-fatal cerebral stroke
Proportion of patients with COVID-19 cases during follow-up | 3 years
  COVID-19 cases during follow-up
Hospitalization due to cardiovascular diseases | 3 years
  Proportion of patients with hospitalization due to cardiovascular diseases
COVID-19-related hospitalization | 3 years
  Pproportion of patients with COVID-19-related hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Republican Scientific and Practical Center of Cardiology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided
Protection of personal data